CLINICAL TRIAL: NCT06427083
Title: An Anonymized, De-identified Registry Study to Determine the Effectiveness and Safety of Weight Loss With Enavogliflozin in Patients With Type 2 Diabetes Mellitus
Brief Title: Registry Study to Determine the Effectiveness and Safety of Weight Loss With Enavogliflozin in Patients With Type 2 Diabetes Mellitus
Status: Active, not recruiting | Type: Observational
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Other Study IDs: DW_ODNENV_DB_02
Record Dates: First submitted 2024-05-14; First posted 2024-05-23 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patient diagnosed with type2 diabetes mellitus: patient diagnosed with type2 diabetes mellitus
  Interventions: Drug: Envlo Tablet; Drug: Envolomet SR Tablet

INTERVENTIONS:
Drug: Envlo Tablet — Enavogliflozin 0.3mg
Drug: Envolomet SR Tablet — Enavogliflozin 0.3mg/Metformin1,000mg

SUMMARY:
This observational study is designed to assess the effects of Envlo Tablet or Envlomet SR Tablet on weight loss and safety in patients with Type 2 diabetes, conducted in real primary care settings over a period of 24 weeks.

DETAILED DESCRIPTION:
The study plans to recruit patients with Type 2 diabetes who are scheduled to receive Envlo Tablet or Envlomet SR Tablet based on the attending physician's medical judgment, regardless of previous diabetes treatment. However, voluntary consent from patients is required for participation in the study, even if Envlo Tablet or Envlomet SR Tablet are prescribed.

Data collection will occur for up to 24 weeks post-Envlo Tablet or Envlomet SR Tablet initiation, capturing demographic information, physical measurements, vital signs, and lifestyle factors. Follow-up visits at 12 weeks and 24 weeks post-baseline will be conducted to collect data, including clinical indicators, safety evaluations, and adverse events. Data will be collected based on routine clinical records, with no mandatory study-specific visits or interventions.

Overall, this observational study aims to collect data on demographics, physical measurements, vital signs, and clinical indicators in patients receiving Envlo Tablet or Envlomet SR Tablet in real-world clinical settings, utilizing information obtained during routine patient care processes.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 19 to 80 years.
2. Patients with Type 2 diabetes who are scheduled to receive initial treatment with Enavogliflozin or Enavogliflozin Extended-Release Tablets based on the attending physician's medical judgment, within the following insurance coverage ranges:

   * Enavogliflozin monotherapy
   * Combination therapy of Enavogliflozin with two agents (metformin)
   * Combination therapy of Enavogliflozin with three agents (metformin + DPP-4 inhibitor)
3. Patients with obesity beyond the pre-obesity stage according to the 2022 Korean Endocrine Society obesity treatment guidelines:

   * Pre-obesity stage: BMI 23~24.9 kg/m2
   * Stage 1 obesity: BMI 25~29.9 kg/m2
   * Stage 2 obesity: BMI 30~34.9 kg/m2
   * Stage 3 obesity: BMI ≥ 35 kg/m2
4. Individuals planning to undertake appropriate exercise and dietary therapy for glycemic control during the observational study period.
5. Fertile women and men who agree to contraception according to appropriate contraceptive methods during the observational study period or have no plans for pregnancy, adhering to methods such as hormonal contraceptives, intrauterine devices or systems, tubal ligation, vasectomy, dual contraception methods (such as cervical cap and male condom), etc.
6. Individuals who have received detailed explanation and have understood the nature of the observational study and the investigational drug, and have provided written consent to participate voluntarily in the observational study and to comply with subject precautions during the study period.

Exclusion Criteria:

1. Individuals with diabetes other than Type 2 diabetes (Type 1 diabetes, diabetic ketoacidosis, gestational diabetes, etc.).
2. Individuals contraindicated for Enavogliflozin or Enavogliflozin Extended-Release Tablets based on the approved indications:

   * Patients with a history of hypersensitivity reactions to the components of Enavogliflozin or Enavogliflozin Extended-Release Tablets
   * Patients with an eGFR (estimated Glomerular Filtration Rate) less than 30 mL/min/1.73m2, end-stage renal disease, or undergoing dialysis
   * Patients with moderate to severe hepatic impairment (AST or ALT > 3 times the upper limit of normal, Total Bilirubin > 2 times the upper limit of normal, hepatitis or hepatic failure)
   * Patients classified as NYHA (New York Heart Association) class III or IV
3. Patients initiating treatment with Enavogliflozin or Enavogliflozin Extended-Release Tablets at enrollment with an eGFR of less than 60 mL/min/1.73m2.
4. Patients with unstable weight due to treatment with obesity drugs or weight loss medications within 3 months prior to enrollment or other treatments (surgery, dietary therapy, etc.).
5. Individuals with diminished mental capacity.
6. Pregnant and lactating women.
7. Individuals currently participating in another clinical trial and receiving investigational drugs or investigational medical devices.
8. Other individuals deemed unsuitable for participation in the observational study based on the investigator's (attending physician's) judgment.

Ages: 19 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The mean and standard deviation of the change from baseline to 12 or 24 weeks in weight and body mass index (BMI) from previously conducted Phase 2 and Phase 3 clinical trials were used as references for calculation using G*Power 3.1.9.7.
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2024-06-11 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
change in BMI | 24 weeks
  change in BMI at 24 weeks from baseline
change in body weight | 24 weeks
  change in body weight at 24 weeks from baseline

SECONDARY OUTCOMES:
change in BMI | 12 weeks
  change in BMI at 12 weeks from baseline
change in body weight | 12 weeks
  change in body weight at 12 weeks from baseline
Proportion of subjects achieving ≥ 5% reduction in BMI | 12 weeks
  Proportion of subjects achieving ≥ 5% reduction in BMI at 12 weeks compared to baseline
Proportion of subjects achieving ≥ 5% reduction in BMI | 24 weeks
  Proportion of subjects achieving ≥ 5% reduction in BMI at 24 weeks compared to baseline
Proportion of subjects achieving ≥ 5% reduction in weight | 12 weeks
  Proportion of subjects achieving ≥ 5% reduction in weight at 12 weeks compared to baseline
Proportion of subjects achieving ≥ 5% reduction in weight | 24 weeks
  Proportion of subjects achieving ≥ 5% reduction in weight at 24 weeks compared to baseline
Change in body composition analyzer indicators (body fat mass, visceral fat mass, muscle mass, waist/hip circumference, etc.) | 12 weeks
  Change in body composition analyzer indicators (body fat mass, visceral fat mass, muscle mass, waist/hip circumference, etc.) at 12 weeks compared to baseline
Change in body composition analyzer indicators (body fat mass, visceral fat mass, muscle mass, waist/hip circumference, etc.) | 24 weeks
  Change in body composition analyzer indicators (body fat mass, visceral fat mass, muscle mass, waist/hip circumference, etc.) at 24 weeks compared to baseline
Change in HbA1c | 12 weeks
  Change in HbA1c at 12 weeks compared to baseline
Change in HbA1c | 24 weeks
  Change in HbA1c at 24 weeks compared to baseline
Change in FPG | 12 weeks
  Change in FPG at 12 weeks compared to baseline
Change in FPG | 24 weeks
  Change in FPG at 24 weeks compared to baseline
Proportion of subjects achieving HbA1c < 7% | 12 weeks
  Proportion of subjects achieving HbA1c < 7% at 12 weeks compared to baseline
Proportion of subjects achieving HbA1c < 7% | 24 weeks
  Proportion of subjects achieving HbA1c < 7% at 24 weeks compared to baseline
Proportion of subjects achieving HbA1c < 6.5% | 12 weeks
  Proportion of subjects achieving HbA1c < 6.5% at 12 weeks compared to baseline
Proportion of subjects achieving HbA1c < 6.5% | 24 week
  Proportion of subjects achieving HbA1c < 6.5% at 24 weeks compared to baseline
Proportion of subjects achieving therapeutic response [change in HbA1c (baseline HbA1c - HbA1c at each evaluation time point) > 0.5% or HbA1c < 7%] | 12 weeks
  Proportion of subjects achieving therapeutic response [change in HbA1c (baseline HbA1c - HbA1c at each evaluation time point) > 0.5% or HbA1c < 7%] at 12 weeks compared to baseline
Proportion of subjects achieving therapeutic response [change in HbA1c (baseline HbA1c - HbA1c at each evaluation time point) > 0.5% or HbA1c < 7%] | 24 weeks
  Proportion of subjects achieving therapeutic response [change in HbA1c (baseline HbA1c - HbA1c at each evaluation time point) > 0.5% or HbA1c < 7%] at 24 weeks compared to baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Kyung Hee University Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided